CLINICAL TRIAL: NCT00052520
Title: Phase I/II Study of Adoptive Immunotherapy With CD8+ WT1-Specific CTL Clones for Patients With Advanced MDS, CML, AML or ALL After Allogeneic Hematopoietic Stem Cell Transplant
Brief Title: Biological Therapy in Treating Patients With Advanced Myelodysplastic Syndrome, Acute or Chronic Myeloid Leukemia, or Acute Lymphoblastic Leukemia Who Are Undergoing Stem Cell Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Merav Bar, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1655.00; NCI-2009-01471 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P01CA018029 (NIH)
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2013-07

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); B-cell Adult Acute Lymphoblastic Leukemia; B-cell Childhood Acute Lymphoblastic Leukemia; Childhood Chronic Myelogenous Leukemia; Childhood Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia; Essential Thrombocythemia; Polycythemia Vera; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Refractory Anemia With Excess Blasts; Refractory Anemia With Excess Blasts in Transformation; Relapsing Chronic Myelogenous Leukemia; Secondary Acute Myeloid Leukemia; T-cell Adult Acute Lymphoblastic Leukemia; T-cell Childhood Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Congenital Abnormalities; Leukemia, Myelomonocytic, Chronic; Thrombocythemia, Essential; Polycythemia Vera; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts | interventions — aldesleukin; Interleukin-2; Peripheral Blood Stem Cell Transplantation; Transplantation; Gene Expression Profiling; Immunologic Techniques; Flow Cytometry; Polymerase Chain Reaction; Cytogenetic Analysis; Coloring Agents; Staining and Labeling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): See Detailed Description
  Interventions: Biological: therapeutic allogeneic lymphocytes; Biological: aldesleukin; Procedure: peripheral blood stem cell transplantation; Procedure: allogeneic bone marrow transplantation; Other: laboratory biomarker analysis; Genetic: gene expression analysis; Other: immunologic technique; Other: flow cytometry; Genetic: polymerase chain reaction; Genetic: cytogenetic analysis; Other: staining method

INTERVENTIONS:
Biological: therapeutic allogeneic lymphocytes — Given IV
  Other Names: ALLOLYMPH
Biological: aldesleukin — Given SC
  Other Names: IL-2; Proleukin; recombinant human interleukin-2; recombinant interleukin-2
Procedure: peripheral blood stem cell transplantation — Undergo transplantation
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Procedure: allogeneic bone marrow transplantation — Undergo transplantation
  Other Names: bone marrow therapy, allogeneic; bone marrow therapy, allogenic; transplantation, allogeneic bone marrow; transplantation, allogenic bone marrow
Other: laboratory biomarker analysis — Correlative studies
Genetic: gene expression analysis — Correlative studies
Other: immunologic technique — Correlative studies
  Other Names: immunological laboratory methods; laboratory methods, immunological
Other: flow cytometry — Correlative studies
Genetic: polymerase chain reaction — Correlative studies
  Other Names: PCR
Genetic: cytogenetic analysis — Correlative studies
Other: staining method — Correlative studies
  Other Names: Staining

SUMMARY:
This phase I/II trial is studying the side effects of biological therapy and to see how well it works in treating patients with advanced myelodysplastic syndrome, chronic myeloid leukemia, acute myeloid leukemia, or acute lymphoblastic leukemia. Biological therapies, including immunotherapy, can potentially be used to stimulate the immune system and stop cancer cells from growing. Immunotherapy given to patients who have undergone donor stem cell transplantation may be a way to eradicate remaining cancer cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and potential toxicities associated with infusing donor CD8+ cytotoxic T lymphocyte (CTL) clones specific for Wilms' tumor (WT1) in patients who have relapsed or at a high risk of relapse post transplant for myelodysplastic syndromes (MDS), chronic myelogenous leukemia (CML), acute myeloid leukemia (AML), or acute lymphoblastic leukemia (ALL).

SECONDARY OBJECTIVES:

I. To determine the in vivo persistence of transferred T cells and assess migration to the bone marrow, a predominant site of leukemic relapse.

II. To determine if adoptively transferred WT1-specific T cells mediate antileukemic activity.

OUTLINE: Donors undergo leukapheresis for stem cell harvest to generate CD8-positive WT1 gene-specific CTL clones at the time of allogeneic stem cell transplantation.

After post-transplantation hematopoietic recovery, patients receive treatment for either highest-risk disease (prophylactically) or relapsed disease.

Highest-risk disease group: Patients receive CD8-positive WT1 gene-specific CTL clones intravenously (IV) over 1-2 hours on days 0, 14, and 28. Beginning 2-4 hours after CTL infusion, patients receive interleukin-2 subcutaneously (SC) twice daily on days 28-42 in the absence of unacceptable toxicity.

Relapsed-disease group: Some patients with evidence of leukemic relapse may receive standard salvage chemotherapy prior to donor CTL infusions and then receive CD8-positive WT1 gene-specific CTL clones and interleukin-2 as in the highest-risk group.

Patients in both groups who have progressive disease after complete or partial response to therapy may be eligible for retreatment with CD8-positive WT1 gene-specific CTL clones.

After completion of study treatment, patients are followed every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility for Enrollment:

  * a.

    * i) Pre-transplant: Patients undergoing allogeneic hematopoietic stem cell transplantation for refractory anemia with excess blasts (RAEB), refractory anemia with excess blasts in transformation (RAEB-t), CML beyond chronic phase, AML beyond first remission, Philadelphia chromosome (BCR-ABL)-positive ALL at any stage, any ALL beyond first remission, primary refractory AML or ALL, therapy-related AML at any stage, or acute leukemia at any stage arising in a patient with an antecedent diagnosis of a myelodysplastic or myeloproliferative syndrome (including chronic myelomonocytic leukemia, CML, polycythemia vera, essential thrombocytosis, and agnogenic myeloid metaplasia with myelofibrosis);
    * ii) Post-transplant: Patients who have relapsed after transplant (morphologic, flow cytometric, cytogenetic and molecular relapse) can be offered enrollment on the protocol and may undergo therapy if it is considered possible to control their disease while waiting for the generation of study therapy
  * b. Patients and donors must both express an human leukocyte antigen (HLA)-allele for which it is possible to generate WT1-specific clones for
  * c. Patients must be able to provide blood and bone marrow samples required for this protocol
* Eligibility for Prophylactic Treatment with CD8+ CTL After Transplant (Highest Risk Subgroup): At time of planned treatment, CD8+ CTL specific for WT1 must have been generated and have completed Quality Control (QC) testing

  * a. Patients must have had > 5% morphologic blasts detectable in bone marrow or peripheral blood just prior to or at the time of transplant
  * b. Patients must have evidence of post transplant recovery of normal hematopoiesis (absolute neutrophil count [ANC] > 500/mm^3) for at least 7 days prior to the initiation of CTL infusions
  * c. Patients on immunosuppressive therapy for graft-versus-host disease (GVHD) are eligible for treatment if not receiving corticosteroids or if the dose of corticosteroids can be tapered to =< the equivalent of 0.5 mg/kg/day of prednisone; the patient's symptoms have to remain stable and unlikely to increase to stage III or IV acute GVHD or chronic GVHD is unlikely to progress following the change in immunosuppressive therapy, after an appropriate monitoring period, as deemed by the patients treating physician and the principal investigator
* Eligibility for Treatment with CD8+ CTL at the Time of Relapse after Transplant (All Others): At time of planned treatment, CD8+ CTL specific for WT1 must have been generated and have completed Quality Control (QC) testing

  * a. Patients must have evidence of recurrent disease post transplant; this includes patients with the following:

    * i) Morphologic relapse defined as one or more of the following: Abnormal peripheral blasts in absence of growth factor therapy; abnormal bone marrow blasts > 5% of nucleated cells; extramedullary chloroma or granulocytic sarcoma
    * ii) Flow cytometric relapse defined as: the appearance in the peripheral blood or bone marrow of cells with an abnormal; immunophenotype detected by flow cytometry that is consistent with leukemia recurrence
    * iii) Cytogenetic relapse defined as: the appearance in one or more metaphases from bone marrow or peripheral blood cells of either a non-constitutional cytogenetic abnormality identified in at least one cytogenetic study performed prior to transplant or a new abnormality known to be associated with leukemia; (for CML) an increase in the number of Ph+ metaphases from bone marrow or peripheral blood between two consecutive samples after engraftment, or; an increase in the percentage of BCR/ABL+ cells by fluorescence in situ hybridization (FISH) between two consecutive samples after engraftment
    * iv) Molecular relapse defined as: one or more positive polymerase chain reaction (PCR) assays for the presence of clonotypic immunoglobulin heavy chain (IgH) or T cell receptor (TCR) gene rearrangement in patients transplanted for B-or T-cell acute lymphoblastic leukemia, respectively; one or more positive post transplant reverse transcription (RT)-PCR assays for the presence of BCR-ABL messenger ribonucleic acid (mRNA) fusion transcripts in patients transplanted for Philadelphia chromosome (BCRABL)-positive acute lymphoblastic leukemia; (for CML) a PCR assay of bone marrow (BM) or peripheral blood mononuclear cell (PBMC) positive for the presence of the BCR/ABL mRNA fusion transcript that quantitatively increases by greater than one order of magnitude on a subsequent sample
  * b. Patients on immunosuppressive therapy for GVHD at the time of relapse are eligible for treatment if not receiving corticosteroids or if the dose of corticosteroids can be tapered to < the equivalent of 0.5 mg/kg/day of prednisone; the patient's symptoms have to remain stable and unlikely to increase to stage III or IV acute GVHD or chronic GVHD is unlikely to progress following the change in immunosuppressive therapy, after an appropriate monitoring period, as deemed by the patients treating physician and the principal investigator
* DONOR: Both the patient and donor must have an HLA-allele which it is possible to generate WT1-specific clones for
* DONOR: If a separate leukapheresis via peripheral intravenous access can be arranged, the stem cell donor will undergo leukapheresis to provide the required PBMC no sooner than 2 weeks before or after the stem cell mobilization and harvest
* DONOR: If a separate leukapheresis is not possible, a portion of the PBMC from the donor's peripheral blood stem cell harvest may potentially be used to generate WT1-specific CTL clones; the feasibility of this option will depend upon the minimal cell dose required for transplantation and the presence of an excess harvest yield and the possibility of generating CTL from this product
* DONOR: Some donors will be asked to provide both a separate leukapheresis and a portion of the peripheral blood mononuclear cells (PBMC) from the donor's peripheral blood stem cell harvest
* DONOR: Leukapheresis donors must be age 18 or older

Exclusion Criteria:

* Patients for whom CD8+ CTL clones specific for WT1 have not been generated in time for planned infusion (these patients can potentially be treated later if CTL become available); Also we will exclude patients whose malignant cells do not over express WT-1, based on direct analysis of a bone marrow sample with > 50% blasts or of leukemia cells isolated for expression analysis; in either case patients will be informed about the availability of other treatment protocols for which they might be eligible
* Patients with Karnofsky performance status or Lansky play score =< 30%
* Patients with current stage III or IV GVHD unresponsive to therapy or requiring therapy with anti-CD3 mAb, prednisone > 0.5 mg/kg/day (or corticosteroid equivalent), or other treatments resulting in the ablation or inactivation of T cells (such as other anti-T cell monoclonal antibodies); although the concurrent use of cyclosporine, FK506, or MMF is not strictly an exclusion criteria, attempts should be made to discontinue it if possible
* Patients requiring concurrent therapy with hydroxyurea or other agents that may interfere with the function or survival of infused CTL clones
* Patients with a preexisting nonhematopoietic organ toxicity that is deemed by the principal investigator to place the patient at unacceptable risk for treatment on the protocol
* Patients with graft rejection or failure
* DONOR: Medical conditions precluding either leukapheresis or blood donation may include but are not limited to:

  * Inadequate age or weight (leukapheresis donors must be age 18 or older, other criteria per physician discretion)
  * Active infection, with or without antibiotic treatment
  * Recent hepatitis exposure, hepatitis A or B antigenemia, or hepatitis C antibody positivity
  * Pregnancy or nursing; HIV or human T-lymphotropic virus (HTLV) infection
  * Severe cardiovascular disease (e.g., uncontrolled hypertension, recent myocardial infarction [MI], or unstable angina)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2002-09; Primary Completion 2011-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Toxicity rate associated with infusing donor CD8+ CTL clones specific for WT1 in patients at high risk for post transplant relapse of CML, AML, or ALL | Up to 4 weeks after the final dose of CTL
  Assessed by Common Terminology Criteria (CTC) version 3.0.

SECONDARY OUTCOMES:
Relapse of disease | Up to 2 years
  Patients achieving complete remission with chemotherapy and T cell infusions will be followed to determine the duration of response. The proportion of responders will be estimated with associated confidence intervals. Duration of remission will be summarized using time-to-event methods, which will allow estimates to be made while some patients remain in remission.

CONTACTS AND LOCATIONS:
Overall Officials: Merav Bar, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States